CLINICAL TRIAL: NCT02539407
Title: Population Pharmacokinetics and Rationalization of Anti-infectives Administration in Critically Ill Children
Brief Title: Population Pharmacokinetics of Anti-infectives in Critically Ill Children
Acronym: OPTIMOME
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-01-08
Record Dates: First submitted 2015-07-02; First posted 2015-09-03 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Pediatric Intensive Care Unit; Pediatric Immuno-hematology Department
Keywords: β-lactam antibiotics; Children; Anti-infectives; Aminoglycosides, glycopeptides; Fluoroquinolone; Fungal; Antiviral
MeSH Terms: interventions — Pharmacokinetics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Anti-infectives: Anti-infectives of the following : β-lactam antibiotics, Aminoglycosides, Glycopeptides, Fluoroquinolone, Daptomycin, Rifampin, Trimethoprim, Sulfamethoxazole, Clarithromycin, Fungal, Antiviral
  Pharmacokinetics
  Interventions: Other: Pharmacokinetics

INTERVENTIONS:
Other: Pharmacokinetics

SUMMARY:
Concentrations and effects of anti-infectives in critically ill children are unpredictable and the risk of under-exposure may be associated with poor clinical outcomes. In addition, between-subject variability (BSV) is known to be substantial in critically ill children. Rationalisation of anti-infectives in children is therefore desirable.

The investigators aim to investigate, using a population approach, the pharmacokinetics (PK) and pharmacodynamics (PD) of anti-infectives including PK/PD targets (fT(%) > minimal inhibitory concentration (MIC)) and PD endpoints (clinical outcomes) in critically ill children. Covariates The effects of covariates on anti-infectives PK and PK/PDs are investigated in order to better explain the BSV and to ultimately suggest individualized dosage regimens.

It will be a prospective PK study including 11 anti-infectives antibiotics. Six blood samples were taken from each patient during dosing interval. The primary PK/ PD targets were anti-infectives concentrations above the MIC of the pathogen at both 50% (50% f T>MIC) and 100% (100% f T>MIC) of the dosing interval. The investigators used skewed logistic regression to describe the effect of anti-infectives exposure on patient outcome.

DETAILED DESCRIPTION:
Background and aims of the study:

Recent studies have suggested a risk of under-exposure to anti-infectives in critically ill adults. This under-exposure may be associated with poor clinical outcomes as well as a delay or incomplete clinical resolution of infection; The dosing regimen of anti-infectives in critically ill children is usually based on weight (i.e. mg per Kg). However, between-subject variability is known to be substantial in children and even more so in critical illness; As a result, concentrations and effects of anti-infectives are unpredictable and the risk of under- or over-exposure is thus genuine and considerable. Rationalisation of anti-infectives in children is therefore desirable.

The purpose of the present study is to investigate, using a population approach, the pharmacokinetics (PK) and pharmacodynamics (PD) of intravenous anti-infectives including usual PK/PD targets (fT(%) > minimal inhibitory concentration (MIC)) and PD endpoints (clinical outcomes) in critically ill children. The effects of developmental and other factors related to critical illness on anti-infectives PK and PK/PDs are investigated in order to better explain the observed between-subject variabilities and to ultimately suggest individualized dosage regimens.

This prospective study will be conducted in six paediatric services of Public Hospitals in Paris, France

Intervention:

Patient selection will take place in the 6 paediatric services. The senior physician proposes the study to holders of parental authority whose child receives or will receive anti-infectives during its follow-up or hospitalization.

The senior physician will give a briefing note to the holders of parental authority, and if the child is able to understand the information. The non-oral opposition for the retrieval and analysis of data will be collected.

No intervention or no charge will be made for this study.

ELIGIBILITY:
Inclusion Criteria:

* Minor patient requiring the administration of an anti-infective belonging to the following classes : β-lactam antibiotics; aminoglycosides, glycopeptides; fluoroquinolones; other antibiotics (daptomycin, rifampin, trimethoprim, sulfamethoxazole, clarithromycin); fungal; antivirals, during its follow-up or hospitalization

Exclusion Criteria:

* Patient and parents having notified to the doctor that they refuse data recovery.

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Minor patients requiring the administration of anti-infectives
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2015-09-11 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
anti-infectives concentration | until 28 days

SECONDARY OUTCOMES:
number of identified or suspected pathogen | until 28 days
composite measure of the health condition | until 28 days
  Clinical data: anthropometric characteristics, organs function, severity score, clinical cure
predictive variables of underdosing/overdosing of antiinfectives and biological evolution | until 28 days
  Clinical data: anthropometric characteristics, organs function, severity score, clinical cure

CONTACTS AND LOCATIONS:
Overall Officials: Oualha Mehdi, MD,PhD, Principal Investigator — Hospital Necker - Enfants Malades; Jean-Marc Treluyer, MD, PhD, Study Chair — EA08 Paris Descartes Pharmacologie et Evaluation des thérapeutiques chez l'enfant et la femme enceinte
Locations (1):
- Hospital Necker - Enfants Malades (Public Hospitals of Paris), Paris, France

REFERENCES:
- [Derived] Berthaud R, Urien S, Krid S, Foissac F, Oualha M, Thy M, Boyer O, Beranger A, Hirt D, Benaboud S, Treluyer J-M, Bouazza N. Cefazolin population pharmacokinetics in children undergoing maintenance hemodialysis for kidney failure. Antimicrob Agents Chemother. 2025 Nov 5;69(11):e0045125. doi: 10.1128/aac.00451-25. Epub 2025 Oct 2. PMID 41036866
- [Derived] Marsaux A, Leger PL, Rambaud J, Bille E, Renolleau S, Treluyer JM, Gana I, Lorrot M, Grimaud M, Toubiana J, Beranger A, Benaboud S, Oualha M. Beta-Lactam Antibiotic Exposure During Pediatric Extracorporeal Membrane Oxygenation: Retrospective Cohort Analysis of Drug Levels Using Standard Dosing, 2018-2020. Pediatr Crit Care Med. 2024 Dec 1;25(12):1127-1137. doi: 10.1097/PCC.0000000000003605. Epub 2024 Oct 7. PMID 39630067
- [Derived] Collignon C, de Marcellus C, Oualha M, Neuranter V, Heilbronner C, Hirt D. Pharmacokinetic profile of acyclovir in a child receiving continuous kidney replacement therapy for acute liver failure. Pediatr Nephrol. 2023 Oct;38(10):3493-3497. doi: 10.1007/s00467-023-05881-6. Epub 2023 Jan 27. PMID 36702934
- [Derived] de Cacqueray N, Boujaafar S, Bille E, Moulin F, Gana I, Benaboud S, Hirt D, Beranger A, Toubiana J, Renolleau S, Treluyer JM, Oualha M. Therapeutic Drug Monitoring of Antibiotics in Critically Ill Children: An Observational Study in a Pediatric Intensive Care Unit. Ther Drug Monit. 2022 Apr 1;44(2):319-327. doi: 10.1097/FTD.0000000000000918. PMID 35292609
- [Derived] Nguyen T, Oualha M, Briand C, Bendavid M, Beranger A, Benaboud S, Treluyer JM, Zheng Y, Foissac F, Winter S, Gana I, Boujaafar S, Lopez V, Berthaud R, Demir Z, Bouazza N, Hirt D. Population Pharmacokinetics of Intravenous Ganciclovir and Oral Valganciclovir in a Pediatric Population To Optimize Dosing Regimens. Antimicrob Agents Chemother. 2021 Feb 17;65(3):e02254-20. doi: 10.1128/AAC.02254-20. Print 2021 Feb 17. PMID 33318012
- [Derived] Abdalla S, Briand C, Oualha M, Bendavid M, Beranger A, Benaboud S, Treluyer JM, Zheng Y, Capito C, Demir Z, Foissac F, Winter S, Gana I, Boujaafar S, Bouazza N, Hirt D. Population Pharmacokinetics of Intravenous and Oral Acyclovir and Oral Valacyclovir in Pediatric Population To Optimize Dosing Regimens. Antimicrob Agents Chemother. 2020 Nov 17;64(12):e01426-20. doi: 10.1128/AAC.01426-20. Print 2020 Nov 17. PMID 32988829
- [Derived] Beranger A, Benaboud S, Urien S, Moulin F, Bille E, Lesage F, Zheng Y, Genuini M, Gana I, Renolleau S, Hirt D, Treluyer JM, Oualha M. Piperacillin Population Pharmacokinetics and Dosing Regimen Optimization in Critically Ill Children with Normal and Augmented Renal Clearance. Clin Pharmacokinet. 2019 Feb;58(2):223-233. doi: 10.1007/s40262-018-0682-1. PMID 29862466
- [Derived] Beranger A, Oualha M, Urien S, Genuini M, Renolleau S, Aboura R, Hirt D, Heilbronner C, Toubiana J, Treluyer JM, Benaboud S. Population Pharmacokinetic Model to Optimize Cefotaxime Dosing Regimen in Critically Ill Children. Clin Pharmacokinet. 2018 Jul;57(7):867-875. doi: 10.1007/s40262-017-0602-9. PMID 28980166